CLINICAL TRIAL: NCT06910969
Title: Multi-Site Randomized Controlled Trial of A Multidisciplinary Intervention for Adults With Chronic Graft Versus Host Disease
Brief Title: Multidisciplinary Intervention for Adults With Chronic Graft-versus-host Disease
Acronym: HORIZONS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Miami Sylvester Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-651
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Bone Marrow Transplant Complications; Graft-versus-Host Disease
Keywords: neoplasms; hematologic diseases; neoplasms by site; hematologic neoplasms; graft-versus-host disease
MeSH Terms: conditions — Graft vs Host Disease; Neoplasms; Hematologic Diseases; Neoplasms by Site; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HORIZONS intervention (Experimental): Participants randomized to HORIZONS plus usual care will complete the following:
  * Questionnaires at baseline, and weeks 10 and 18
  * Receive the HORIZONS intervention from enrollment and for up to 8 weeks. HORIZONS is an 8-session multidisciplinary, patient-centered intervention that combines medical and psychosocial expertise to enhance self-management and quality of life.
  * Receive usual care as determined by their local clinicians
  Interventions: Behavioral: HORIZONS Intervention
- Minimally enhanced usual care (Active Comparator): Participants randomized to usual care will complete the following
  * Questionnaires at baseline, and weeks 10 and 18 after enrollment
  * Receive a standardized booklet containing evidence-based information on chronic GVHD management and HCT survivorship recommendations as well as receive care as determined by their local oncologists
  Interventions: Behavioral: Minimally enhanced usual care

INTERVENTIONS:
Behavioral: HORIZONS Intervention — Therapist-delivered multidisciplinary group-based telehealth intervention comprised of 8 sessions
  Arms: HORIZONS intervention
Behavioral: Minimally enhanced usual care — Receiving a standardized booklet with evidence-based information on chronic GHVD management and HST survivorship recommendations
  Arms: Minimally enhanced usual care

SUMMARY:
The goal of this study is to demonstrate the efficacy of a multidisciplinary group-based telehealth intervention (HORIZONS) compared to minimally enhanced usual care for improving self-management and quality of life for hematopoietic stem cell transplant (HSCT) survivors living with chronic graft-versus host disease, and to identify critical facilitators and barriers for HORIZONS implementation and adoption.

DETAILED DESCRIPTION:
This is a randomized clinical trial to determine whether a multidisciplinary group-based telehealth intervention is effective at improving the quality of life and reducing psychosocial distress in patients living with chronic graft-versus-host disease. The HORIZONS intervention was developed with the goal of improving the experience and needs of patients living with chronic graft-versus-host disease.

Participants will be randomized into one of the two study groups: HORIZONS plus usual care or minimally enhanced usual care.

Participation in this study is expected to last up to 18 weeks after enrollment.

The investigators expect that about 350 adult allogeneic hematopoietic cell transplant recipients with moderate to severe chronic graft versus host disease will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) who have undergone allogeneic HCT
* Have moderate to severe cGVHD based on patient-report
* Have ability to participate in English or Spanish language group telehealth intervention.

Exclusion Criteria:

* Patients with mild cGVHD based on their self-report.
* Patients with a major untreated psychiatric or cognitive condition which the treating oncology clinicians believes interferes with the capacity to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Patient quality of life (QOL) as measured by the Functional Assessment of Cancer Therapy-BMT (FACT-BMT) questionnaire | 10 weeks
  Compare patient QOL as measured by the FACT-BMT between the two study groups. The FACT-BMT ranges from 0-164 with higher scores indicating better QOL

SECONDARY OUTCOMES:
Patient quality of life (QOL) as measured by the Functional Assessment of Cancer Therapy-BMT (FACT-BMT) questionnaire | Up to 18 weeks post enrollment
  Compare patient QOL as measured by the FACT-BMT between the two study groups. The FACT-BMT ranges from 0-164 with higher scores indicating better QOL
Patient depression symptoms as measured by the Hospital Anxiety and Depression Scale (HADS-Depression) | Up to 18 weeks post enrollment
  Compare depression symptoms as measured by the HADS-Depression between the study groups. The HADS-Depression ranges from 0-21 with higher scores indicating worse depression symptoms
Patient anxiety symptoms as measured by the Hospital Anxiety and Depression Scale (HADS-Depression) | Up to 18 weeks post enrollment
  Compare anxiety symptoms as measured by the HADS-Anxiety between the study groups. The HADS-Anxiety ranges from 0-21 with higher scores indicating worse depression symptoms.
Patient chronic graft-versus-host disease symptoms as measured with the Lee Symptom Scale | Up to 18 weeks post enrollment
  Compare chronic graft versus host disease symptoms as measured by the Lee Symptom Scale. The Lee Symptom Scale ranges from 0 -100 with higher scores indicating worse symptomatology

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Areej El-Jawahri (ael-jawahri@mgb.org). The protocol and statistical analysis plan will be made available on Clinicaltrials.gov as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation